CLINICAL TRIAL: NCT05494749
Title: Effectiveness Of Zirconia Reinforced Glass Ionomer Used In Alternative Restorative Treatment In Molar Incisor Hypomineralization (A Randomized Controlled Clinical Trial And Finite Element Analysis)
Brief Title: Zirconia Reinforced Glass Ionomer in MIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIH_2022
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: zirconomer
- Control (Active Comparator)
  Interventions: Other: HVGI-Equia Forte

INTERVENTIONS:
Other: zirconomer — teeth meeting the inclusion criteria are assigned to receive Zirconomer® restorations
  Arms: Test group
Other: HVGI-Equia Forte — teeth meeting the inclusion criteria are assigned to receive HVGI-Equia Forte® restorations.
  Arms: Control

SUMMARY:
Molar-incisor hypomineralization (MIH) is a qualitative enamel defect, in which molars and incisors involved are prone to post-eruptive enamel breakdown leading to sensitivity, and caries. Atraumatic/Alternative Restorative Treatment (ART) is a minimally invasive procedure. It can be very beneficial in managing MIH-affected molars in communities with limited access to dental care. Zirconia-reinforced GI was recently introduced. It is claimed to serve as a long-term temporary restoration until a more permanent restoration is placed

ELIGIBILITY:
Inclusion Criteria:

* Children free from any systemic disease (ASA I).
* Cooperative children showing positive or definitely positive behavior according to Frankl rating scale
* Hypomineralized first permanent molars that are restorable according to MIH Treatment Need Index (MIH-TNI): Index (2a), (2b), (4a), (4b)
* Teeth with dentinal lesions corresponding to ICDAS II score 5 or 6
* No clinical or radiographic evidence of pulpal involvement.

Exclusion Criteria:

* Index (0), (1), (2c), (3), (4c) on the MIH Treatment Need Index.
* Patients whose parents will not give their consent to participate in the study
* Non-restorable first permanent molars indicated for extraction

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in clinical success rate | at 3 months, 6 months, 9 months, 12 months
  It will be assessed using Modified ART criteria, restorations receiving a score of:
  (0) Restoration is present and satisfactory OR
  (1) Restoration is present, slight defect at the cavity margin of less than 0.5 mm; no repair is needed.
  will be considered successful, and any other score will be considered a failure.

SECONDARY OUTCOMES:
Change in pain | at 1 week, 3 months, 6 months, 9 months, 12 months
  Pain will be recorded using VAS Using a visual analog scale (VAS), the subjects were instructed how to point to the position of the line between faces to indicate how much painthey might feel. In this system, the total scores range from 0 to 100 based on measuring the distance in millimeters from the left end bar to the mark made by the child on the 10 cm line anchored by happy to sad faces, with a higher score indicating more severe pain.
Change in sensitivity | at 1 week, 3 months, 6 months, 9 months, 12 months
  sensitivity will be recorded using VAS by performing air blast test Using a visual analog scale (VAS), the subjects were instructed how to point to the position of the line between faces to indicate how much pain they might feel. In this system, the total scores range from 0 to 100 based on measuring the distance in millimeters from the left end bar to the mark made by the child on the 10 cm line anchored by happy to sad faces, with a higher score indicating more severe pain.
Finite element analysis | 12 months
  Performance of both Zirconomer and HVGI-Equia Forte under dynamic occlusal loads will be assessed using Finite Element Analysis using ANSYS software.

CONTACTS AND LOCATIONS:
Overall Officials: Reham A Mahfouz, MSc, Principal Investigator — Alexandria University, Faculty of Dentistry
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt

REFERENCES:
- [Derived] Mahfouz RA, Hanno AG, Rahman AMAE. Zirconia-reinforced glass ionomer restorations in molar incisor hypomineralization: a randomized controlled clinical trial. Clin Oral Investig. 2025 May 8;29(6):290. doi: 10.1007/s00784-025-06352-y. PMID 40335753